CLINICAL TRIAL: NCT04534829
Title: Efficacy of Fluoroscopic Versus Ultrasound Guided Sacroiliac Joint Radiofrequency Ablation: A Randomized Control Trial
Brief Title: Fluoroscopic vs Ultrasound Guided Sacroiliac (SI) Joint Radiofrequency Ablation
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study cancelled
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00102343
Record Dates: First submitted 2020-07-20; First posted 2020-09-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Sacroiliac Joint Somatic Dysfunction
Keywords: Radiofrequency Ablation; Fluoroscopy; Ultrasound; Sacroiliac joint
MeSH Terms: interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Intervention Model Description: Patients who present with pain thought to be originating from the SIJ will be screened for study participation with fluoroscopy-guided sacral lateral branch blocks (LBB). If a patient has an initial successful sacral LBB (defined as 70% reduction in pain), or has prior successful SIJ RFA, they will be approached for consent to be contacted for study participation. Upon obtaining written consent for study participation, patients will be randomized into one of two groups; US-guided SIJ RFA or fluoroscopy-guided SIJ RFA (current gold-standard). Upon being randomized to either group they will then undergo a second confirmatory sacral LBB under their respective image guidance to confirm candidacy for RFA. If this second, confirmatory LBB is successful (70% pain relief) they qualify for RFA. Then, SIJ RFA will be performed under each respective imaging modality and patients will be followed to document pain improvement, functional outcomes, quality of life and medication use for 18 months.
Who Masked: Outcomes Assessor
Masking Description: In terms of blinding, the principal investigators will be blinded to which arm each study participant is randomized to. It is not possible to blind study participants, as they will be aware of the imaging modality used to perform the procedure. The clinicians serving as private investigators (one in each study arm) will not be blinded to the procedure they are performing. Therefore, this is a single-blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided SIJ RFA (Experimental): Utilizing short axis views, the S1, S2 and S3 foramen and tubercles would be localized and marked by a surgical skin marker. Then, the ultrasound transducer will be moved laterally to achieve a long axis view between the S1 and S2 tubercle. Local skin and subcutaneous tissue freezing would be performed with Lidocaine 1% utilizing a 30-gauge needle. An 18-gauge radiofrequency (RF) cannula will be directed utilizing an in-plane approach toward the S2 and S3 lateral branches between the S2 and S3 tubercles. A small amount of 1% lidocaine will be injected in order to provide comfort.
  The RF generator will be set to continuous monopolar RF ablation and the needle will be heated to 80 degrees Celsius for 90 seconds. The needle will then be repositioned proximally to obtain a slightly larger burn in a similar fashion previously described. A similar approach will be utilized for the S1 lateral branch RF ablation between the S1 and S2 tubercles.
  Interventions: Procedure: Ultrasound-guided Radiofrequency Ablation
- Fluoroscopic-Guided SIJ RFA (Active Comparator): An anterior-posterior approach is used to identify the S1-S3 foramen. A 3-inch spinal needle would be used for marking. Local tissue freezing would be accomplished with Lidocaine 1% and a 30-G needle. An 18-G RF cannula will be positioned over the 12 o'clock position of the S1 foramen and a second cannula placed in the 2 o'clock or 10 o'clock position for the right and left respectively (4-5 mm distance between the cannula). A small amount of 1% lidocaine will be injected for comfort. A lateral projection is taken to ensure the needles are not placed into the foramen. The RF generator will be set to continuous bipolar RF ablation and heated to 80 degrees Celsius for 90 seconds. Then another 18-G RF cannula will be positioned at the 4 o'clock or 8 o'clock position (4-5 mm distance between the cannula) to achieve the second RF ablation. The third RF ablation will be performed with the RF cannula at the 6 o'clock position. An identical fashion is utilized at the S2 and S3 foramen.
  Interventions: Procedure: Fluoroscopic-guided Radiofrequency Ablation

INTERVENTIONS:
Procedure: Fluoroscopic-guided Radiofrequency Ablation — Radiofrequency ablation of the posterior SIJ complex under fluoroscopic-guidance
  Arms: Fluoroscopic-Guided SIJ RFA
Procedure: Ultrasound-guided Radiofrequency Ablation — Radiofrequency ablation of the posterior SIJ complex under ultrasound-guidance
  Arms: Ultrasound-Guided SIJ RFA

SUMMARY:
The sacroiliac joint (SIJ) is estimated to be the source of low mechanical back pain in 10-27% of patients. When conservative measures for treating SIJ pain fail (physiotherapy, exercise, analgesic medications, chiropractic manipulation, etc.) radiofrequency ablation (RFA) is a treatment option in carefully selected patients. RFA uses a radiofrequency generator to create a thermal lesion, with the aim of ablating the nerves that innervate the SIJ complex. Studies have confirmed that SIJ RFA can provide significant relief for patients with SIJ pain. The current gold standard is the use of fluoroscopic (x-ray guidance) to visualize bony landmarks in order to create an accurate thermal lesion along the lateral sacral crest; where the nerves that innervate the SIJ complex reside. Recent literature has proposed a technique for an ultrasound-guided approach to achieve an RFA lesion in patients with SIJ pain. It is proposed that with ultrasound-guidance, versus fluoroscopic-guidance, the interventionalist is able to perform fewer needle passes for the procedure, as well as fewer thermal lesions, thereby achieving shorter performance times. The proposed study serves as a non-inferiority randomized controlled trial to assess the effectiveness of ultrasound-guided versus fluoroscopy-guided RFA for the treatment of SIJ pain.

DETAILED DESCRIPTION:
Current practice for SIJ pain that is refractory to conservative treatment, is the use of RFA of the posterior sacral network under fluoroscopic-guidance. There is high variability regarding the long-term benefits of this procedure. To date, there have been no clinical studies evaluating the effectiveness of US-guided RFA procedures for SIJ pain. A study performed in 2017 attempted to determine the effectiveness of US-guided sacral LBBs compared to fluoroscopic-guidance (gold standard in current practice). The results were in favour of an US-guided approach. Compared with fluoroscopy, US-guided sacral lateral branch blocks required a shorter performance time, fewer needle passes, and was associated with a lower incidence of vascular breach. Furthermore, with an US-guided procedure, the patient is no longer exposed to ionizing radiation.With an improved understanding of SIJ sensory innervation, as well as technical improvements in RFA electrodes, it is postulated that RFA under ultrasound-guidance will lead to non-inferior clinical outcomes, as well as shorter performance time and reduced costs compared with the current practice of fluoroscopic-guidance.

The objectives of the current study are the following:

1. To evaluate the efficacy of US-guided posterior sacral network SIJ RFA compared to fluoroscopy-guided SIJ RFA.
2. To compare the post-procedure pain/flare-up and duration required to achieve full recovery for each approach.
3. To perform a cost effectiveness analysis comparing ultrasound and fluoroscopy-guided SIJ RFA.
4. To determine the safety of US-guided SIJ RFA by tracking intra-operative and post-procedure complications.

Research Method/Procedures:

The proposed study is a single-blind, single-center randomized controlled trial. Patients who present with pain thought to be originating from the SIJ will be screened for study participation with fluoroscopy-guided sacral LBBs. If a patient has an initial successful sacral LBB (defined as 70% reduction in pain), or has prior successful SIJ RFA, they will be approached for consent to be contacted for study participation by a member of the HealthPointe team; specifically, patients who consent to be contacted for study participation, will have their charts reviewed by independent assessors for inclusion and exclusion criteria. If a patient meets the inclusion criteria (listed below), they will be contacted by a HealthPointe team member, specifically a nurse or care manager, for study participation. If the patient expresses an interest with the initial contact, they will be subsequently contacted by a study sub-investigator.

Upon obtaining written consent for study participation, patients will be randomized into one of two groups; US-guided SIJ RFA or fluoroscopy-guided SIJ RFA (current gold-standard). Upon being randomized to either group they will then undergo a second confirmatory sacral LBB under their respective image guidance to confirm candidacy for RFA. If this second, confirmatory LBB is successful (70% pain relief or more) the patient qualifies for RFA. Then, SIJ RFA will be performed under each respective imaging modality and patients will be followed to document pain improvement, functional outcomes, quality of life and medication use for 18 months. Study participants will be asked to perform a daily VAS pain diary for the first 6 weeks post-procedure in order to document post-procedure pain flare. Questionnaires will be administered either in person (if appropriate), or by email or over the phone, at 6 weeks, 12 weeks, 6 months, 12 months and 18 months post-RFA procedure.

The primary endpoint is 12 months post-procedure, however the investigators plan to follow for 18 months to determine long-term effectiveness. The investigators will perform an interim-analysis at the 6-month follow-up time period.

In further analyses, the effect of the intervention groups on secondary outcomes listed below will be evaluated:

The average time (in days) for post-procedure pain flare. Pain medication use post-procedure (% increase or decrease from baseline). Participation in physiotherapy and exercise programs (as a binary variable: yes or no) Cost effectiveness analysis comparing procedures based on the following mean data: performance time, radiation time, number of thermal lesions performed, number of RFA needle passes, volume of local anesthetic used. Cost will be compared based on mean data for fluoroscopy- and ultrasound-guided procedures, as well as the cost of monopolar vs. bipolar RFA.

Safety: this will include intra-operative complications related directly to the intervention, as well as post-operative complications and adverse events over the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Body Mass Index (BMI) ≤35
* Clinical presentation must be in keeping with SIJ pain based on both history (pain below L5 vertebrae, localized to the SIJ area, back pain greater than leg pain) and/or physical examination (≥2/5 SIJ provocative tests).
* Diagnosis confirmed by having >70% index pain relief with fluoroscopy-guided SIJ lateral branch blocks (with local anesthetic). Participants will require confirmatory lateral branch block under their respective image modality once randomized, requiring >70% pain relief for diagnosis, prior to completing the randomized SIJ RFA procedure.

Exclusion Criteria:

* Age <18
* Pregnant or inadequate birth control methods (to prevent the exposure of a pregnant female and/or fetus to radiation).
* Inflammatory spondyloarthropathy
* Fibromyalgia
* Radiculopathy (will require an electromyography study to rule out radiculopathy if clinically suspected in patients with primarily buttock pain)
* Discogenic low mechanical back pain
* Symptomatic spinal stenosis
* Generalized or local infection
* Coagulopathy
* Allergy to local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Pain reduction: change from baseline pain scores | 6 weeks to 18 months post-procedure.
  Visual analog scale (VAS) for pain at the various follow-up time periods. The visual analog scale is a numerical scale from 0 to 10; with 0 representing no pain and 10 representing the worst pain imaginable.
Function and quality of life | 6 weeks to 18 months post-procedure.
  Pain, Disability and Quality of Life Questionnaire- Spine (PDQQ-S)

SECONDARY OUTCOMES:
Post-procedure pain flare | Daily visual analog scale (VAS) for pain for the first 6 weeks.
  Daily visual analog scale (VAS) for pain for the first 6 weeks post-procedure to document post-procedure pain flare. The visual analog scale is a numerical scale from 0 to 10; with 0 representing no pain and 10 representing the worst pain imaginable.
Pain medication usage | 6 weeks to 18 months post-procedure.
  Percentage increase or decrease from patients baseline.
Cost effectiveness | Costs compared based on procedural data upon study completion, an average of 18 months.
  Compare study arms based on the following mean data; performance time, radiation time, number of thermal lesions performed, number of RFA needle passes, volume of local anesthetic used. Cost will be compared based on mean data for fluoroscopy- and ultrasound-guided procedures, as well as the cost of monopolar vs. bipolar RFA

OTHER OUTCOMES:
Participation in physical therapy | 6 weeks to 18 months post-procedure.
  Binary variable (yes/no) to document confounding data.

CONTACTS AND LOCATIONS:
Overall Officials: Shane Hoeber, M.D., Principal Investigator — University of Alberta
Locations (1):
- HealthPointe, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aydin SM, Gharibo CG, Mehnert M, Stitik TP. The role of radiofrequency ablation for sacroiliac joint pain: a meta-analysis. PM R. 2010 Sep;2(9):842-51. doi: 10.1016/j.pmrj.2010.03.035. PMID 20869684
- [Background] Cohen SP, Chen Y, Neufeld NJ. Sacroiliac joint pain: a comprehensive review of epidemiology, diagnosis and treatment. Expert Rev Neurother. 2013 Jan;13(1):99-116. doi: 10.1586/ern.12.148. PMID 23253394
- [Background] Dreyfuss P, Henning T, Malladi N, Goldstein B, Bogduk N. The ability of multi-site, multi-depth sacral lateral branch blocks to anesthetize the sacroiliac joint complex. Pain Med. 2009 May-Jun;10(4):679-88. doi: 10.1111/j.1526-4637.2009.00631.x. PMID 19638143
- [Background] Finlayson RJ, Etheridge JB, Elgueta MF, Thonnagith A, De Villiers F, Nelems B, Tran DQ. A Randomized Comparison Between Ultrasound- and Fluoroscopy-Guided Sacral Lateral Branch Blocks. Reg Anesth Pain Med. 2017 May/Jun;42(3):400-406. doi: 10.1097/AAP.0000000000000569. PMID 28178092
- [Background] Roberts SL, Burnham RS, Ravichandiran K, Agur AM, Loh EY. Cadaveric study of sacroiliac joint innervation: implications for diagnostic blocks and radiofrequency ablation. Reg Anesth Pain Med. 2014 Nov-Dec;39(6):456-64. doi: 10.1097/AAP.0000000000000156. PMID 25304483
- [Background] Roberts SL, Burnham RS, Agur AM, Loh EY. A Cadaveric Study Evaluating the Feasibility of an Ultrasound-Guided Diagnostic Block and Radiofrequency Ablation Technique for Sacroiliac Joint Pain. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):69-74. doi: 10.1097/AAP.0000000000000515. PMID 27811527
- [Background] Roberts SL, Stout A, Loh EY, Swain N, Dreyfuss P, Agur AM. Anatomical Comparison of Radiofrequency Ablation Techniques for Sacroiliac Joint Pain. Pain Med. 2018 Oct 1;19(10):1924-1943. doi: 10.1093/pm/pnx329. PMID 29415262